CLINICAL TRIAL: NCT04161222
Title: Effectiveness of Specific Core Activation Protocol on Lower Limb Stability in Soccer Players
Brief Title: Effectiveness of a Protocol of Specific Activation.
Acronym: Knee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cadiz (Other)
Responsible Party: Principal Investigator, Manuel Rodriguez Huguet, Clinical Professor, University of Cadiz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cádiz CF
Record Dates: First submitted 2019-11-05; First posted 2019-11-13 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Injuries:Knee Injuries
Keywords: Knee stability.; Core; Gluteus medius; Warm-up; Football
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: A specialist physician will be diagnosed the process.
Who Masked: Participant
Masking Description: Outcomes assesor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The control group will perform a typical warm-up of competitive football, added to a specific activation of gluteus medius and core.
  Interventions: Other: Experimental group
- Control group (Experimental): The control group will perform a typical warm-up of competitive football.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Experimental group — Experimental group will perform a typical warm-up of competitive football, added to a specific activation of gluteus medius and core.
  Arms: Experimental group
Other: Control group — Control group will perform a typical warm-up of competitive football
  Arms: Control group

SUMMARY:
In football, knee is the joint that suffers the most severe injuries. Sometimes, this is produced by poor pre-activation of the musculature that is responsible for knee stability and central stability.

OBJETIVE: Study the efficacy of specific gluteus medius and core activation protocol in knee stability in youth football players.

DETAILED DESCRIPTION:
A randomized, longitudinal clinical trial with a blinded and prospective evaluator will be carried out, in which the knee stability will be evaluated with the following tests: Y-balance test and Flamingo balance test. The measurements will be made before and after the intervention. The study will be carried out with patients evaluated by a specialist in Traumatology and will be randomly divided by a system of numerical tables through a computer program between the experimental and control groups. The control group will perform a typical warm-up of competitive football; and the experimental one will do this above, added to a specific activation of gluteus medius and core. Dynamic stability (Y-balance test) and postural and static stability (Flamingo balance test) will be measured before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Perform soccer sports practice, at least 3 times a week at a competitive level.

Exclusion Criteria:

* Subjects with a knee surgery.
* Patients who are injured at the time of the study.

Ages: 18 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Y-balance test | Baseline
  Y-balance test Measures the strength of the lower limb, neuromuscular control, flexibility and dynamic balance

SECONDARY OUTCOMES:
Y-balance test | Baseline and four weeks.
  Y-balance test Measures the strength of the lower limb, neuromuscular control, flexibility and dynamic balance.
Flamingobalance test | Baseline and four weeks.
  Flamingo balance test measures postural balance and static balance.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Rodriguez Huguet, Study Director — University of Cádiz
Locations (1):
- Ciudad Deportiva Bahía de Cádiz, Puerto Real, Cádiz, Spain

REFERENCES:
- [Background] Ekstrand J, Walden M, Hagglund M. A congested football calendar and the wellbeing of players: correlation between match exposure of European footballers before the World Cup 2002 and their injuries and performances during that World Cup. Br J Sports Med. 2004 Aug;38(4):493-7. doi: 10.1136/bjsm.2003.009134. PMID 15273193
- [Background] Rahnama N, Reilly T, Lees A. Injury risk associated with playing actions during competitive soccer. Br J Sports Med. 2002 Oct;36(5):354-9. doi: 10.1136/bjsm.36.5.354. PMID 12351333
- [Background] Falese L, Della Valle P, Federico B. Epidemiology of football (soccer) injuries in the 2012/2013 and 2013/2014 seasons of the Italian Serie A. Res Sports Med. 2016 Oct-Dec;24(4):426-432. doi: 10.1080/15438627.2016.1239105. Epub 2016 Sep 29. PMID 27683952
- [Background] Peterson L, Junge A, Chomiak J, Graf-Baumann T, Dvorak J. Incidence of football injuries and complaints in different age groups and skill-level groups. Am J Sports Med. 2000;28(5 Suppl):S51-7. doi: 10.1177/28.suppl_5.s-51. PMID 11032108
- [Background] Alentorn-Geli E, Myer GD, Silvers HJ, Samitier G, Romero D, Lazaro-Haro C, Cugat R. Prevention of non-contact anterior cruciate ligament injuries in soccer players. Part 1: Mechanisms of injury and underlying risk factors. Knee Surg Sports Traumatol Arthrosc. 2009 Jul;17(7):705-29. doi: 10.1007/s00167-009-0813-1. Epub 2009 May 19. PMID 19452139
- [Background] Zazulak BT, Hewett TE, Reeves NP, Goldberg B, Cholewicki J. Deficits in neuromuscular control of the trunk predict knee injury risk: a prospective biomechanical-epidemiologic study. Am J Sports Med. 2007 Jul;35(7):1123-30. doi: 10.1177/0363546507301585. Epub 2007 Apr 27. PMID 17468378
- [Background] Nguyen AD, Shultz SJ, Schmitz RJ, Luecht RM, Perrin DH. A preliminary multifactorial approach describing the relationships among lower extremity alignment, hip muscle activation, and lower extremity joint excursion. J Athl Train. 2011 May-Jun;46(3):246-56. doi: 10.4085/1062-6050-46.3.246. PMID 21669093
- [Background] Zazulak BT, Hewett TE, Reeves NP, Goldberg B, Cholewicki J. The effects of core proprioception on knee injury: a prospective biomechanical-epidemiological study. Am J Sports Med. 2007 Mar;35(3):368-73. doi: 10.1177/0363546506297909. Epub 2007 Jan 31. PMID 17267766
- [Background] Huxel Bliven KC, Anderson BE. Core stability training for injury prevention. Sports Health. 2013 Nov;5(6):514-22. doi: 10.1177/1941738113481200. PMID 24427426
- [Background] Dello Iacono A, Padulo J, Ayalon M. Core stability training on lower limb balance strength. J Sports Sci. 2016;34(7):671-8. doi: 10.1080/02640414.2015.1068437. Epub 2015 Jul 15. PMID 26177151
- [Background] Leetun DT, Ireland ML, Willson JD, Ballantyne BT, Davis IM. Core stability measures as risk factors for lower extremity injury in athletes. Med Sci Sports Exerc. 2004 Jun;36(6):926-34. doi: 10.1249/01.mss.0000128145.75199.c3. PMID 15179160
- [Background] Panjabi MM. The stabilizing system of the spine. Part I. Function, dysfunction, adaptation, and enhancement. J Spinal Disord. 1992 Dec;5(4):383-9; discussion 397. doi: 10.1097/00002517-199212000-00001. PMID 1490034
- [Background] Akuthota V, Nadler SF. Core strengthening. Arch Phys Med Rehabil. 2004 Mar;85(3 Suppl 1):S86-92. doi: 10.1053/j.apmr.2003.12.005. PMID 15034861
- [Background] Liemohn WP, Baumgartner TA, Gagnon LH. Measuring core stability. J Strength Cond Res. 2005 Aug;19(3):583-6. doi: 10.1519/1533-4287(2005)19[583:MCS]2.0.CO;2. PMID 16095406
- [Background] Haruyama K, Kawakami M, Otsuka T. Effect of Core Stability Training on Trunk Function, Standing Balance, and Mobility in Stroke Patients. Neurorehabil Neural Repair. 2017 Mar;31(3):240-249. doi: 10.1177/1545968316675431. Epub 2016 Nov 9. PMID 27821673
- [Background] Escamilla RF, Lewis C, Bell D, Bramblet G, Daffron J, Lambert S, Pecson A, Imamura R, Paulos L, Andrews JR. Core muscle activation during Swiss ball and traditional abdominal exercises. J Orthop Sports Phys Ther. 2010 May;40(5):265-76. doi: 10.2519/jospt.2010.3073. PMID 20436242
- [Background] Borghuis J, Hof AL, Lemmink KA. The importance of sensory-motor control in providing core stability: implications for measurement and training. Sports Med. 2008;38(11):893-916. doi: 10.2165/00007256-200838110-00002. PMID 18937521
- [Background] Eickmeyer SM. Anatomy and Physiology of the Pelvic Floor. Phys Med Rehabil Clin N Am. 2017 Aug;28(3):455-460. doi: 10.1016/j.pmr.2017.03.003. Epub 2017 May 27. PMID 28676358
- [Background] Zhou D, Zhang S, Zhang H, Jiang L, Zhang J, Fang J. A Novel Method of Evaluating Knee Joint Stability of Patients with Knee Osteoarthritis: Multiscale Entropy Analysis with A Knee-Aiming Task. Sci Rep. 2017 Mar 23;7(1):354. doi: 10.1038/s41598-017-00411-5. PMID 28336915
- [Background] Cervenka JJ, Decker MN, Ruhde LA, Beaty JD, Ricard MD. Strength and Stability Analysis of Rehabilitated Anterior Cruciate Ligament Individuals. Int J Exerc Sci. 2018 Jun 1;11(1):817-826. doi: 10.70252/MUNO4563. eCollection 2018. PMID 29997727